CLINICAL TRIAL: NCT05711394
Title: A Phase 3, Multicenter, 12-Week, Double Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of Atogepant for the Preventive Treatment of Episodic Migraine in Pediatric Subjects 6-17 Years of Age.
Brief Title: A Study to Assess the Adverse Events and Change in Disease Activity of Oral Atogepant Tablets in Pediatric Participants (6-17 Years of Age) With Episodic Migraine
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: M21-201; 2022-501100-94-00 (Other: EU CT)
Record Dates: First submitted 2023-01-26; First posted 2023-02-03 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Episodic Migraine
Keywords: Episodic Migraine; Atogepant; QULIPTA; AGN-241689
MeSH Terms: interventions — atogepant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Open-Label PK Substudy: Atogepant Dose A (6-11 yrs) (Experimental): Participants aged 6 to 11 will receive oral tablets of atogepant Dose A to determine appropriate dose for the 6-11 year old group in double-blind treatment period.
  Interventions: Drug: Atogepant
- Open-Label PK Substudy: Atogepant Dose B (6-11 yrs) (Experimental): Participants aged 6 to 11 will receive oral tablets of atogepant Dose B to determine appropriate dose for the 6-11 year old group in double-blind treatment period.
  Interventions: Drug: Atogepant
- Double-Blind Treatment Period: High Dose Atogepant (12-17 yrs) (Experimental): Participants aged 12 to 17 will receive oral tablets of high dose atogepant once a day for 12 weeks.
  Interventions: Drug: Atogepant
- Double-Blind Treatment Period: Placebo (12-17 yrs) (Placebo Comparator): Participants aged 12 to 17 will receive oral tablets of placebo-matching atogepant once a day for 12 weeks.
  Interventions: Drug: Placebo-Matching Atogepant
- Double-Blind Treatment Period: Low Dose Atogepant (12-17 yrs) (Experimental): Participants aged 12 to 17 will receive oral tablets of low dose atogepant once a day for 12 weeks.
  Interventions: Drug: Atogepant
- Double-Blind Treatment Period: High Dose Atogepant (6-11 yrs) (Experimental): Participants aged 6-11 will receive oral tablets of high dose atogepant once a day for 12 weeks.
  Interventions: Drug: Atogepant
- Double-Blind Treatment Period: Placebo (6-11 yrs) (Placebo Comparator): Participants aged 6 to 11 will receive oral tablets of placebo-matching atogepant once a day for 12 weeks.
  Interventions: Drug: Placebo-Matching Atogepant
- Double-Blind Treatment Period: Low Dose Atogepant (6-11 yrs) (Experimental): Participants aged 6-11 will receive oral tablets of low dose atogepant once a day for 12 weeks.
  Interventions: Drug: Atogepant

INTERVENTIONS:
Drug: Atogepant — Oral Tablet
  Other Names: QULIPTA; AGN-241689
  Arms: Double-Blind Treatment Period: High Dose Atogepant (12-17 yrs); Double-Blind Treatment Period: High Dose Atogepant (6-11 yrs); Double-Blind Treatment Period: Low Dose Atogepant (12-17 yrs); Double-Blind Treatment Period: Low Dose Atogepant (6-11 yrs); Open-Label PK Substudy: Atogepant Dose A (6-11 yrs); Open-Label PK Substudy: Atogepant Dose B (6-11 yrs)
Drug: Placebo-Matching Atogepant — Oral Tablet
  Arms: Double-Blind Treatment Period: Placebo (12-17 yrs); Double-Blind Treatment Period: Placebo (6-11 yrs)

SUMMARY:
A migraine is a moderate to severe headache on one side of the head. A migraine attack is a headache that may be accompanied by throbbing, nausea, vomiting, sensitivity to light and sound, or other symptoms. A number of treatments are available for adults with migraine but there are limited approved treatments available for pediatric participants. The main goal of the study is to evaluate the safety and efficacy (how well treatment works) of a low-dose and high-dose of atogepant in pediatric participants between the ages of 6 and 17.

Atogepant is a medicine currently approved to treat adults with migraine (0 to 14 migraine days per month) and is being studied in pediatric participants between the ages of 6 and 17 with a history of episodic migraine. This is a Phase 3, randomized, double-blind study of atogepant in participants with a history of episodic migraine with an open-label pharmacokinetic substudy. Eligible participants will be randomized into 6 different groups. Participants between the ages of 12 and 17 will be randomized to receive placebo, low-dose atogepant, or high-dose atogepant for 12 weeks. Participants between the ages of 6 and 11 will also be randomized to receive placebo, low-dose atogepant, or high-dose atogepant for 12 weeks. The specific atogepant doses to be used in participants between the ages of 6 and 11 will be determined after the PK substudy is complete. Around 450 participants will be enrolled in approximately 100 sites worldwide.

Placebo, low-dose atogepant, and high-dose atogepant are given as a tablet to take by mouth once a day. At the end of Week 12, participants will either undergo a follow-up visit 4 weeks after last study treatment or join an extension study where they can continue to receive atogepant for another 52 weeks.

There may be a bigger responsibility for participants in this study. Participants will attend regular visits during the study at a hospital or clinic. The effects of treatment will be checked by medical assessments, blood tests, checking for side effects, and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Weight is >= 20 kg (44 lbs) and < 135 kg (298 lbs).
* History of episodic migraine with or without aura consistent with a diagnosis according to the International Classification of Headache Disorders (ICHD) -3 (2018) for at least 6 months.
* Participant has to have 4 to 14 migraine days and < 15 headache days in the 28-day baseline period per eDiary.
* To be eligible for the PK substudy, participants must be 6 to 11 years of age (inclusive), with a history of migraine (consistent with a diagnosis according to the ICHD-3 [2018]) and per investigator judgment is appropriate to receive preventive treatment for migraine.

Exclusion Criteria:

* History of migraine brainstem aura, hemiplegic migraine, or retinal migraine as defined by ICHD-3 (2018).
* Have a current diagnosis of chronic migraine as defined by ICHD-3 (2018).
* Have a current diagnosis of new daily persistent headache, trigeminal autonomic cephalgia (e.g., cluster headache), or painful cranial neuropathy as defined by ICHD-3 (2018).

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 450 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Mean Monthly Migraine Days | Baseline (Week 0) through Week 12
  A migraine day is defined as any calendar day on which a migraine occurs as per participant eDiary. Calendar days begin at midnight and last until 11:59 PM.
Number of Participants Experiencing Adverse Events | Baseline (Week 0) through Week 16
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Change from Baseline in Mean Monthly Headache Days | Baseline (Week 0) through Week 12
  A headache day is defined as any calendar day on which headache pain lasting 2 hours or longer occurs unless an acute headache medication (e.g., ibuprofen, triptan) was used after the start of the headache, in which case no minimum duration will be specified. Calendar days begin at midnight and last until 11:59 PM.
Change from Baseline in Mean Monthly Headache Days of at Least Moderate Severity | Baseline (Week 0) through Week 12
  A headache day is defined as any calendar day on which headache pain lasting 2 hours or longer occurs unless an acute headache medication (e.g., ibuprofen, triptan) was used after the start of the headache, in which case no minimum duration will be specified. Calendar days begin at midnight and last until 11:59 PM.
Change from Baseline in Mean Monthly Acute Medication Use Days | Baseline (Week 0) through Week 12
  An acute medication use day is defined as any day on which a participant reports, per eDiary, the intake of allowed medication(s) for the acute treatment of migraine.
Percentage of Participants who Achieve at least a 50% Reduction in Average of Monthly Migraine Days | Baseline (Week 0) to 3 Months
  A migraine day is defined as any calendar day on which a migraine occurs as per participant eDiary. Calendar days begin at midnight and last until 11:59 PM.
Change from Baseline in the Pediatric Quality of Life Inventory (PedsQL) total score | Baseline (Week 0) through Week 12
  The PedsQL is a 23-item measure that evaluates quality of life in four areas of functioning: physical, emotional, social, and school functioning. The PedsQL yields a total quality of life score and two summary scores: Physical Health Summary Score and Psychosocial Health Summary Score.
Change from baseline in the Pediatric Migraine Disability Assessment (PedMIDAS) total score | Baseline (Week 0) through Week 12
  The PedMIDAS scale evaluates the impact of headache on school performance, disability at home and social/sport function. The score is a composite of the total of 6 questions.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (98):
- United States (42):
  - Rehabilitation & Neurological Services /ID# 248517, Huntsville, Alabama
  - The Center for Clinical Trials - Saraland /ID# 271604, Saraland, Alabama
  - Preferred Research Partners /ID# 249729, Little Rock, Arkansas
  - Preferred Research Partners /ID# 270406, Little Rock, Arkansas
  - Advanced Research Center /ID# 251381, Anaheim, California
  - Alliance for Research Alliance for Wellness /ID# 248521, Long Beach, California
  - Excell Research, Inc /ID# 247532, Oceanside, California
  - Lumos Clinical Research Center /ID# 249731, San Jose, California
  - Sunwise Clinical Research /ID# 248529, Walnut Creek, California
  - Advanced Neurosciences Research, LLC /ID# 247592, Fort Collins, Colorado
  - Northwest Florida Clinical Research Group, LLC /ID# 251382, Gulf Breeze, Florida
  - Advanced Research Institute of Miami /ID# 248539, Homestead, Florida
  - My Preferred Research LLC /ID# 249720, Miami, Florida
  - Asclepes Research Centers - Spring Hill /ID# 248525, Spring Hill, Florida
  - Coastal Georgia Child Neurology /ID# 249733, Brunswick, Georgia
  - Deaconess Clinic - Gateway Health Center /ID# 247589, Newburgh, Indiana
  - College Park Family Care Center Overland Park /ID# 249734, Overland Park, Kansas
  - Michigan Headache & Neurological Institute (MHNI) /ID# 247468, Ann Arbor, Michigan
  - Proven Endpoints LLC /ID# 258066, Ridgeland, Mississippi
  - Cognitive Clinical Trials (CCT) - Papillion /ID# 248536, Papillion, Nebraska
  - Goryeb Childrens Hospital /ID# 249724, Morristown, New Jersey
  - Dent Neurologic Institute - Amherst /ID# 248534, Amherst, New York
  - Modern Migraine MD /ID# 258074, New York, New York
  - Headache Wellness Center /ID# 251018, Greensboro, North Carolina
  - Patient Priority Clinical Sites, LLC /ID# 247535, Cincinnati, Ohio
  - Cincinnati Childrens Hospital Medical Center /ID# 258070, Cincinnati, Ohio
  - CincyScience /ID# 249726, West Chester, Ohio
  - Lynn Institute of Oklahoma City /ID# 247600, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia - Main /ID# 258071, Philadelphia, Pennsylvania
  - Le Bonheur Children's Hospital /ID# 261084, Memphis, Tennessee
  - Access Clinical Trials, Inc. /ID# 248532, Nashville, Tennessee
  - UT Health Austin at Dell Children's Neurology Clinic /ID# 264082, Austin, Texas
  - FutureSearch Trials of Neurology /ID# 247470, Austin, Texas
  - 3A Research - East El Paso /ID# 248516, El Paso, Texas
  - Earle Research /ID# 248501, Friendswood, Texas
  - Family Psychiatry of The Woodlands /ID# 249727, The Woodlands, Texas
  - ClinPoint Trials /ID# 248540, Waxahachie, Texas
  - Pantheon Clinical Research /ID# 251601, Bountiful, Utah
  - Alpine Research Organization - Clinton /ID# 276497, Clinton, Utah
  - Highland Clinical Research /ID# 247590, Salt Lake City, Utah
  - Office of Maria Ona /ID# 249738, Franklin, Virginia
  - Core Clinical Research /ID# 249721, Everett, Washington
- Belgium (2):
  - Uza /Id# 247339, Edegem, Antwerpen
  - AZ Sint-Jan Brugge /ID# 247201, Bruges, West-Vlaanderen
- Canada (3):
  - Stollery Children's Hospital /ID# 249672, Edmonton, Alberta
  - London Health Sciences Center- University Hospital /ID# 252979, London, Ontario
  - McGill University Health Centre - Glen Site. /ID# 247271, Montreal, Quebec
- Denmark (3):
  - Herlev Hospital /ID# 247724, Herlev, Capital Region
  - Regionshospitalet Godstrup /ID# 247902, Herning, Central Jutland
  - Aalborg Sygehus Nord /ID# 247428, Aalborg, North Denmark
- France (3):
  - CHU Amiens-Picardie Site Sud /ID# 248833, Amiens, Somme
  - Centre Hosp Intercommunal de Creteil /ID# 248832, Créteil, Val-de-Marne
  - CHU Toulouse - Hôpital des enfants /ID# 247553, Toulouse
- Hungary (2):
  - MIND Clinic /ID# 248687, Budapest
  - Semmelweis Egyetem /ID# 248360, Budapest
- Israel (5):
  - Shamir Medical Center /ID# 256857, Beer Ya'akov, Central District
  - Hillel Yaffe Medical Center /ID# 246747, Hadera, Haifa District
  - The Chaim Sheba Medical Center /ID# 246746, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 247466, Tel Aviv, Tel Aviv
  - Bnai Zion Medical Center /ID# 247469, Haifa
- Italy (3):
  - Fondazione IRCCS Istituto Neurologico Carlo Besta /ID# 247581, Milan, Milano
  - Ospedale Pediatrico Bambino Gesù /ID# 247647, Rome, Roma
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone /ID# 247638, Palermo
- Japan (7):
  - Konan Medical Center /ID# 254457, Kobe, Hyōgo
  - Yamaguchi Clinic /ID# 254753, Nishinomiya, Hyōgo
  - Umenotsuji Clinic /ID# 254453, Kochi, Kochi
  - Sendai Headache and Neurology Clinic Medical Corporation /ID# 254211, Sendai, Miyagi
  - Tominaga Clinic - Osaka /ID# 254450, Osaka, Osaka
  - Tokyo Medical University Hospital /ID# 254459, Shinjuku-ku, Tokyo
  - Tatsuoka Neurology Clinic /ID# 254455, Kyoto
- Netherlands (3):
  - Canisius-Wilhelmina Ziekenhuis /ID# 253065, Nijmegen, Gelderland
  - HagaZiekenhuis /ID# 247318, The Hague, South Holland
  - ZorgSaam Zorggroep Zeeuws-Vlaanderen /ID# 247301, Terneuzen, Zeeland
- Poland (6):
  - Clinical Research Center Medic-R /ID# 247383, Poznan, Greater Poland Voivodeship
  - Athleticomed Sp. z o.o /ID# 248789, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Specjalistyczne Gabinety Sp. z o.o. /ID# 247384, Krakow, Lesser Poland Voivodeship
  - Indywidualna Praktyka Lekarska dr hab. med. Anna Szczepanska-Szerej /ID# 247382, Lublin, Lublin Voivodeship
  - OHA-MED sp. z o.o /ID# 248614, Warsaw, Masovian Voivodeship
  - MIGRE Polskie Centrum Leczenia Migreny Anna Gryglas-Dworak /ID# 247381, Wroclaw
- Puerto Rico (5):
  - Clinical Research Investigator Group, LLC /ID# 261254, Bayamón
  - Dr. Samuel Sanchez PSC /ID# 248495, Caguas
  - Puerto Rico Health Institute /ID# 249741, Dorado
  - CMRC Headlands LLC /ID# 251634, San Juan
  - PRCCI Clinical Research Center /ID# 262726, San Juan
- Romania (3):
  - Spitalul Clinic de Copii Dr. Victor Gomoiu /ID# 248431, Bucharest, București
  - Spitalul Clinic de Urgenta pentru Copii Cluj Napoca /ID# 248595, Cluj-Napoca, Cluj
  - Delta Health Care S.R.L /ID# 248130, Bucharest
- Spain (5):
  - Hospital Universitario Vall de Hebron /ID# 247967, Barcelona
  - Hospital Clinico San Carlos /ID# 249267, Madrid
  - Hospital Universitario 12 de Octubre /ID# 275578, Madrid
  - Hospital Universitario Virgen del Rocio /ID# 248632, Seville
  - Hospital Universitario y Politecnico La Fe /ID# 247969, Valencia
- Sweden (2):
  - Sodersjukhuset /ID# 248279, Stockholm, Stockholm County
  - Vastra Gotealandsregionen Regionhalsan /ID# 248277, Mölnlycke
- United Kingdom (4):
  - Great Ormond Street Children's Hospital /ID# 262933, London, Greater London
  - Medway NHS Foundation Trust /ID# 249065, Gillingham, Kent
  - NHS Grampian /ID# 249067, Aberdeen
  - Stepping Hill Hospital-Stockport NHS foundation trust /ID# 261121, Stockport

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M21-201